CLINICAL TRIAL: NCT03490617
Title: Misoprostol Prior To Cupper Intra Uternine Device Insertion In Nullipara: A Randomized Clinical Trial
Brief Title: Misoprostol Prior to IUD Insertion in Nullipara
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Principal Investigator, Melania Amorim, PhD, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MISO DIU 01
Record Dates: First submitted 2013-03-04; First posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-03

CONDITIONS: Family Planning
Keywords: Intrauterine device; Misoprostol; Nulliparous women; Contraception

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaginal Misoprostol Group (Active Comparator): Vaginal misoprostol (400 μg) 4 hours prior to IUD insertion
  Interventions: Drug: Vaginal misoprostol
- Placebo group (Placebo Comparator): Vaginal placebo tablets 4 hours prior to IUD insertion
  Interventions: Drug: Vaginal misoprostol

INTERVENTIONS:
Drug: Vaginal misoprostol — To determine effectiveness of vaginal misoprostol to facilitate IUD insertion in nulligravida women
  Other Names: Prostokos

SUMMARY:
The use of misoprostol at a dose of 400 µg administered vaginally four hours prior to IUD insertion increased the ease of insertion and reduced the incidence of pain during the procedure, although the frequency of cramps increased following misoprostol use.

DETAILED DESCRIPTION:
Nulligravidas women of reproductive age were submitted to IUD insertion between July 2009 and November 2011 at the Instituto de Medicina Integral Prof. Fernando Figueira in Recife, Pernambuco, Brazil. A total of 179 women were randomly allocated to two groups: 86 to use 400 µg of misoprostol vaginally four hours prior to IUD insertion and 93 to use placebo. Risk ratios (RR) were calculated as measures of relative risk, together with their 95% confidence intervals (95%CI). The number needed to treat (NNT) and the number needed to harm (NNH) were also calculated.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* No chirurgical procedure in the cervix
* Wish to use IUD as a contraceptive method

Exclusion criteria are as follows:

* Presence of active cervical infection visible upon speculum exam (purulent cervicits)
* Pelvic Inflammatory Disease (PID) or other uterine infection diagnosed within the last 3 months (based on self-report or clinical documentation)
* Pregnancy ending less than 6 weeks prior to enrollment in study
* History of prior IUD placement
* History of uterine cavity abnormality including Mullerian tract anomalies and leiomyomas distorting uterine cavity shape
* History of uterine surgery
* Allergy or intolerance to misoprostol or other prostaglandin
* Undiagnosed abnormal vaginal bleeding
* Malignancy of the genital tract
* Allergy to any component of the IUD or Wilson's disease (for copper- containing IUDs)
* Pre-procedure use of anesthesia or analgesia (including use of narcotics, benzodiazepines, or use of anesthetic beyond use at the tenaculum site)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2009-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Cervical dilatation | four hours after misoprostol use
  the frequency of women with cervical dilation ≤ 4 mm (measured by inserting a #4 Hegar dilator through the internal orifice of the cervix uteri immediately prior to IUD insertion

SECONDARY OUTCOMES:
Difficulty in inserting IUD | four hours after misoprostol use
  subjective difficulty (as reported by the investigator) in inserting the IUD and classified as difficult, very difficult and easy
Pain at insertion | four hours after misoprostol use
  judged subjectively by the woman and evaluated by the investigator using a visual analogue scale (VAS). The scale ranged from 0 to 10, in which zero is the absence of pain and 10 the worst pain imaginable.

OTHER OUTCOMES:
Subjective sensation as reported by the woman | four hours after misoprostol use
  the woman's subjective evaluation of the procedure (IUD insertion)was classified as not disagreeable, slightly disagreeable, disagreeable or very disagreeable.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Medicina Integral Professor Fernando Figueira, Recife, Pernambuco, Brazil